CLINICAL TRIAL: NCT07114237
Title: The Effect of Opioid Free Anesthesia in Morbid Obese Patient Undergoing Gynecological Surgeries Using Ultrasound-Guided Bilateral Transversus Abdominus Plane Block and Dexmedetomidine Infusion: A Randomized Controlled
Brief Title: The Effect of Opioid Free Anesthesia Using Ultrasound-Guided Bilateral Transversus Abdominus Plane Block and Dexmedetomidine Infusion
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Merihan Alaa Eldin Ahmed, Resident, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 36264MS694/9/24
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-05

CONDITIONS: Anesthesia; Opioid; Gynecological Surgery
Keywords: Gynecological Surgeries; Opioid Free Anesthesia; Morbid Obese; Dexmedetomidine Infusion
MeSH Terms: interventions — Control Groups; Anesthesia, General

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I: Opioid Free Anesthesia group (Experimental): patients will receive opioid free anesthesia and bilateral ultrasound guided transversus abdominus plane block
  Interventions: Procedure: Opioid Free Anesthesia
- Group II: Control group (Placebo Comparator): patients will receive conventional general anesthesia
  Interventions: Procedure: Control group (general anesthesia)

INTERVENTIONS:
Procedure: Opioid Free Anesthesia — patients will receive opioid free anesthesia and bilateral ultrasound guided transversus abdominus plane block.
  Arms: Group I: Opioid Free Anesthesia group
Procedure: Control group (general anesthesia) — patients will receive conventional general anesthesia
  Arms: Group II: Control group

SUMMARY:
This study aimed to determine the effects of Opioid-free anesthesia using dexmedetomidine and bilateral Transversus abdominis plane block on the quality of recovery, incidence of Opioid-free anesthesia, and post-operative pain and delirium in morbid obese patients undergoing gynecological surgeries.

DETAILED DESCRIPTION:
Opioid analgesic drugs have been the most commonly used perioperative pain-relieving medications for a very long time. While they are effective at relieving somatic pain they, unfortunately, do not eliminate neuropathic pain and have a profound potential for developing addiction.

The most significant opioid side effect is respiratory depression. This is especially important in patients with obesity, sleep apnea, chronic obstructive pulmonary disease and operations that are associated with a high incidence of post-operative respiratory failure.

Opioid may also induce post-operative nausea and vomiting , pruritus, urine retention, postoperative delirium. Furthermore, opioids depress cell mediated immunity and, in some studies, opioids have been found to be associated with an increased tumor recurrence rate after cancer surgery.

Opioid-free anesthesia has become more and more popular among anesthesiologists around the world. It is an emerging technique and a recent research perspective based on the idea that avoiding intraoperative opioids would be associated with better postoperative outcomes. It allows opioid-sparing and better outcomes than morphine administered as a sole analgesic agent after surgery. Opioid-free anesthesia is based on the same concept, as one drug will not replace opioids. It is the association of drugs and/or techniques that allows a good quality general anesthesia with no need for opioids. Dexmedetomidine is an alpha-2 agonist with analgesic action. Unlike opioids it is not associated with significant respiratory depression, post-operative nausea and vomiting, pruritus, constipation, ileus or delirium.

In laparoscopic surgeries, it has been found to provide adequate analgesia when used as the only analgesic. It provides enhanced recovery and patient satisfaction after laparotomy and should be considered as part of any enhanced recovery after surgery program.

Transversus abdominis plane block is a regional anesthesia technique that involves injecting a local anesthetic into the transversus abdominis plane. It is a triangular fascial plane located between the internal oblique (IO) and the transversus abdominis muscles.

This study aimed to determine the effects of Opioid-free anesthesia using dexmedetomidine and bilateral Transversus abdominis plane block on the quality of recovery, incidence of Opioid-free anesthesia, and post-operative pain and delirium in morbid obese patients undergoing gynecological surgeries.

ELIGIBILITY:
Inclusion Criteria:

* 50 female patients aged 21-65 years.
* Patients with a Body mass index≥ 35 kg/m2
* American society of Anesthesiology class II-III.
* Undergoing elective gynecological surgeries.

Exclusion Criteria:

* Patient refusal.
* History of allergy to local anesthetic.
* Liver or renal pathology affecting drug elimination.
* Mental dysfunction or cognitive disorders.
* Patients on chronic pain medications.
* Hypotension, bradycardia, atrioventricular block, intraventricular or sinoatrial block.
* Coagulopathy

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female patients
Enrollment: 150 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
quality of recovery on postoperative day | one day
  The Quality of Recovery-40 questionnaire scores. The Quality of Recovery-40 questionnaire includes five dimensions of recovery: physical comfort (12 items), emotional state (9 items), physical independence (5 items), psychological support (7 items), and pain (7 items).

SECONDARY OUTCOMES:
Postoperative pain severity | 24 HOURS
  Postoperative pain severity will be assessed by the numerical rating scale ( 0 no pain while 10 is the maximum pain).

CONTACTS AND LOCATIONS:
Overall Officials: Merihan Ahmed, Resident, Principal Investigator — Tanta University
Locations (1):
- Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF